CLINICAL TRIAL: NCT04946188
Title: Non-invasive Monitoring to Translate the Biometric Data of Participants With Diabetes Into Blood Glucose Levels
Brief Title: Translating Biometric Data Into Blood Glucose Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scimita Operations Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-02-099
Record Dates: First submitted 2021-04-22; First posted 2021-06-30 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Type 2
Keywords: Non-invasive; Blood Glucose Levels; Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Opuz NICGM (Experimental): Participants will be provided with one non-invasive, custom-built prototype device (study device), which they will use throughout their day-to-day life/activities over the study period.
  Interventions: Device: Opuz NICGM

INTERVENTIONS:
Device: Opuz NICGM — A wearable and non-invasive prototype device that allows for measurement of bioimpedance data with the aim to help develop a mathematical model to predict blood glucose levels.
  Other Names: Opuz Device; Opuz Ring

SUMMARY:
This study is designed to assist with the development of a first, truly non-invasive technology for blood glucose monitoring, which will have the potential to eliminate the need for painful finger pricking or expensive continuous blood glucose monitor use. The purpose of this study is to collect biometric data, such as bioimpedance (how well the body impedes electric current flow), from participants who are living with type 2 diabetes. A proof-of-concept prototype (non-invasive continuous glucose monitor; NI-CGM) will be used to collect this biometric data. The data will then be used to develop and refine a computer model that can be used to predict blood glucose levels (BGLs). Individuals with diabetes experience a great range of blood BGLs throughout their daily life and activities, therefore it is essential to gather biometric data corresponding to this large range to build a computer model, to ensure model reliability.

DETAILED DESCRIPTION:
The study will be conducted over a two-week period where the participants are required to wear the prototype, that will continuously collect the biometric data. Participants are required to use this device together with two existing commercially available blood glucose meters that are considered management routine for diabetes (an Abbott FreeStyle Libre and an Accu-Chek® Mobile), throughout the duration of the study. The majority of the study is carried out independently, by the participants, where they wear the prototype throughout their daily life and activities. The data collected from the non-invasive custom-built device and the existing blood glucose meters will be used to develop a computer model that will allow for blood glucose levels to be predicted, over time.

The study will not interfere with any of the participants' diabetes management plans provided to them, by their regular doctor, under regular care, such as medications, diet and current use of blood glucose monitoring.

It is hypothesised that the bioimoedance data collected using the non-invasive prototype device, in conjunction with existing devices used in diabetes management, will enable the development of a computer model that allows for blood glucose levels to be predicted in people with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 70 years
* Physician diagnosis of Type 2 diabetes
* Haemoglobin A1c (HbA1c) range between 7 - 10%
* Body mass index between 20 - 40
* Regularly eats 3 meals per day (breakfast, lunch, and dinner)
* Technologically literate (e.g. able to use Apps, smart phones)
* Able to commit to attending the Sponsor site
* Able to commit to wearing a non-invasive, custom-built device through most daily activities
* Currently self-monitoring their BGL and able to commit to taking measurements at least 6 times per day
* Proficiency in reading and writing in English

Exclusion Criteria:

* Currently on insulin therapy (other than long-acting insulin therapy)
* Currently pregnant, pregnant in the last 6 months, or planning a pregnancy
* Currently breastfeeding
* Current smoker
* Any other confounding major disease or condition as deemed appropriate by investigator, determined by review of medical history and/or patient reported medical history
* Clinically unstable or rapidly progressing diabetic retinopathy, neuropathy, and/or frequent nausea, bloating or vomiting, sever gastroesophageal reflux, or early satiety.
* Multiple medications (taking more than 10 medications is often an indicator of having multiple major comorbidities which is an exclusion criteria. Furthermore, we want to exclude potential multiple drug interactions with blood glucose levels which may impact results of study)
* Currently on active curative treatments for cancer
* Currently receiving systemic glucocorticoid therapy
* Using lipid-lowering medication at a dose that has not been stable for the past 3 months
* History of reactions to alcohol wipes, antiseptics, or adhesives (isobornyl acrylate which is the adhesive used for attachment of Freestyle Libre sensors and may cause contact dermatitis)
* Using an insulin pump
* Pacemaker fitted
* Fasting C-peptide levels below 0.5 ng/mL or above 2.0 ng/mL
* Has had an episode of diabetic ketoacidosis in the past 6 months
* Has had an episode of severe hypoglycemia within the past 6 months
* Currently unstable blood glucose control
* Receiving dialysis treatment
* Has had a blood transfusion or severe blood loss within the past 3 months
* Unwilling to self-monitor their BGL (at least 6 measurement, daily)
* Currently participating in another clinical study
* Known to the Investigators
* Other investigator-determined criteria making participants unsuitable for participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Generation of a predictive models for determining blood glucose levels | at 14 days post introduction of intervention
  Performance of computer models for blood glucose level estimation using collected bioimpedance spectroscopy data.
Validation of predictive model for determining blood glucose levels | at 14 days post introduction of intervention
  Performance of predictive models will be evaluated using the consensus error grid. Mean Absolute Relative Difference (MARD) and Consensus Error Grid (CEG) distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Telfer, PhD (Med), Principal Investigator — Scimita Operations; Farid Sanai, PhD (Med), Study Chair — Scimita Operations
Locations (1):
- Scimita Operations, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
All data have already gone through a careful process of de-identification. Data can be made available after study completion for the purposes of further research, and to develop and validate the model after quality checks and Secondary analyses. Data will be available to all investigators who provide a sound proposal, as well case-by-case basis at the discretion of Primary Sponsor and PI Dr Thomas Telfer.
Time Frame: De-identified data is expected to be available after study completion and following publication of results, with no determined end date.
Access Criteria: Data obtained from this study will be made available after approval from PI Dr Thomas Telfer.
  Scimita ventures t.telfer@scimitaventures.com
  +61 481848190

REFERENCES:
- [Background] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507
- [Background] Villena Gonzales W, Mobashsher AT, Abbosh A. The Progress of Glucose Monitoring-A Review of Invasive to Minimally and Non-Invasive Techniques, Devices and Sensors. Sensors (Basel). 2019 Feb 15;19(4):800. doi: 10.3390/s19040800. PMID 30781431
- [Background] D. K. Kamat, D. Bagul, and P. M. Patil, "Blood Glucose Measurement Using Bioimpedance Technique," Adv. Electron., vol. 2014, pp. 1-5, 2014, doi: 10.1155/2014/406257
- [Background] Tura A. Noninvasive glycaemia monitoring: background, traditional findings, and novelties in the recent clinical trials. Curr Opin Clin Nutr Metab Care. 2008 Sep;11(5):607-12. doi: 10.1097/MCO.0b013e328309ec3a. PMID 18685457
- [Background] P. Daarani & A.Kavithamani, "Blood glucose level monitoring by noninvasive method using near infra red sensor," Int. J. Latest Trends Eng. Technol., vol. IRES, no. 1, 2017, doi: 10.21172/1.ires.19
- [Background] N. D. Nanayakkara, S. C. Munasingha, and G. P. Ruwanpathirana, "Non-invasive blood glucose monitoring using a hybrid technique," in MERCon 2018 - 4th International Multidisciplinary Moratuwa Engineering Research Conference, pp. 7-12, 2018, doi: 10.1109/MERCon.2018.8421885
- [Background] Ding S, Schumacher M. Sensor Monitoring of Physical Activity to Improve Glucose Management in Diabetic Patients: A Review. Sensors (Basel). 2016 Apr 23;16(4):589. doi: 10.3390/s16040589. PMID 27120602
- [Background] Valensi P, Extramiana F, Lange C, Cailleau M, Haggui A, Maison Blanche P, Tichet J, Balkau B; DESIR Study Group. Influence of blood glucose on heart rate and cardiac autonomic function. The DESIR study. Diabet Med. 2011 Apr;28(4):440-9. doi: 10.1111/j.1464-5491.2010.03222.x. PMID 21204961
- [Background] Mueller M, Talary MS, Falco L, De Feo O, Stahel WA, Caduff A. Data processing for noninvasive continuous glucose monitoring with a multisensor device. J Diabetes Sci Technol. 2011 May 1;5(3):694-702. doi: 10.1177/193229681100500324. PMID 21722585
- See also: World Health Organisation. (2018, Oct. 30). Diabetes — https://www.who.int/news-room/fact-sheets/detail/diabetes

DOCUMENTS (1):
  • Informed Consent Form (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT04946188/ICF_000.pdf